CLINICAL TRIAL: NCT01215890
Title: A Randomized, Data Collection Program To Determine the Efficacy and Safety of Risedronate (Actonel) Therapy Plus Calcium and Vitamin D Supplementation Versus Placebo Plus Calcium and Vitamin D Supplementation in the Treatment of Low Bone Mineral Density in Crohn's Disease Patients
Brief Title: Risedronate Therapy in the Treatment of Low Bone Mineral Density in Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Other Study IDs: RIS-RF
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Crohn's Disease; Low Bone Mineral Density
Keywords: Crohn's disease; Low bone mineral density; inflammatory bowel disease; bisphosphonate
MeSH Terms: conditions — Crohn Disease; Bone Diseases, Metabolic; Inflammatory Bowel Diseases | interventions — Risedronic Acid

ARMS (2):
- risedronate plus calcium and viamin D (Active Comparator)
  Interventions: Drug: risedronate
- placebo plus clacium and vitamin D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: risedronate
  Arms: risedronate plus calcium and viamin D
Drug: placebo
  Arms: placebo plus clacium and vitamin D

SUMMARY:
The occurrence of bone loss in Crohn's disease patients is an important clinical problem for both patients with and without active disease. While therapy does exist for treatment and prevention of low BMD, evidence of its efficacy in Crohn's disease patients is lacking. The current standard of therapy in Canada for the treatment of osteoporosis is etidronate, with adequate calcium and vitamin D supplementation.

The primary objective of the study is to assess the efficacy of risedronate, compared to placebo, administered once-weekly, in the treatment of low BMD of the spine and hip in patients with Crohn's disease at 12 months, based on an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age, or older.
* Crohn's disease, as documented by clinical, radiologic, endoscopic or histologic examination.
* Osteoporosis (T score less than -2.5) or osteopenia (T score between -1.0 and -2.5), as determined by dual energy X-ray absorptiometry.

Exclusion Criteria:

* Known bone disorders other than osteoporosis (such as hyperparathyroidism, Paget's disease, renal osteodystrophy and documented osteomalacia)
* Abnormal thyroid function. Those patients on thyroxine replacement must not have had a change in dose in the two months prior to prospective data collection program entry
* Clinically significant renal impairment (serum creatinine ≥ 2x normal).
* Clinical Short Bowel Syndrome
* Patients on total parenteral or enteral nutrition
* Spinal anatomy that would not allow adequate assessment of lateral spine using DEXA
* Patients who had received:

  1. previous bisphosphonate therapy
  2. fluoride supplement in the 24 months prior to entry
  3. calcium supplements of more than 1.0g/day in the 6 months prior to entry
  4. vitamin D supplements greater than 1000 IU/day in the 6 months prior to entry
  5. calcitonin in the 3 months prior to entry
* Females on hormone replacement therapy who do not agree to continue the therapy for the duration of the prospective data collection program
* Men on testosterone who do not agree to continue it for the duration of the prospective data collection program
* Pregnancy or women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Richard Fedorak, MD, Principal Investigator — University of Alberta
Locations (1):
- Gastrointestinal and Liver Disease Research (GILDR) Group, Edmonton, Alberta, Canada